CLINICAL TRIAL: NCT02018601
Title: Intercostal Nerves Block in the Midaxillary Line Versus Paravertebral Block, Ultrasound Guided Blocks for no Reconstructive Breast Surgery. Randomized Trial
Brief Title: Intercostal Nerves Block in the Midaxillary Line Versus Paravertebral Block for no Reconstructive Breast Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paula Diéguez García (Other)
Responsible Party: Sponsor-Investigator, Paula Diéguez García, anesthesiologist, Complexo Hospitalario Universitario de A Coruña
Organization: Complexo Hospitalario Universitario de A Coruña (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ProsMaMa 13.1
Record Dates: First submitted 2013-12-10; First posted 2013-12-23 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: no Reconstructive Breast Surgery
MeSH Terms: interventions — dexketoprofen trometamol; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BRILMA&dexketoprofen&paracetamol (Experimental): dexketoprofen: 50 mg/8h paracetamol: 1gr/6h
  Interventions: Procedure: BRILMA; Drug: dexketoprofen; Drug: paracetamol
- paravertebral block&dexketoprofen&paracetamol (Active Comparator): dexketoprofen: 50 mg/8h paracetamol: 1g/6h
  Interventions: Procedure: paravertebral block; Drug: dexketoprofen; Drug: paracetamol

INTERVENTIONS:
Procedure: BRILMA
  Other Names: intercostal nerves block in the midaxillary line
  Arms: BRILMA&dexketoprofen&paracetamol
Procedure: paravertebral block
  Arms: paravertebral block&dexketoprofen&paracetamol
Drug: dexketoprofen
Drug: paracetamol

SUMMARY:
The main objectives of the trial are the efficacy and safety of intercostal nerve block in the midaxillary line versus paravertebral block, both guided by ultrasound in patients scheduled for not reconstructive breast surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for not reconstructive unilateral breast surgery.
2. Physical status American Society Anesthesiologists (ASA) I-III.
3. Signed informed consent.
4. Aged between 18 and 75 years.
5. Ability to assess pain using a verbal and numerical scales.
6. Assessment of pain at the time of inclusion in the study is lower than 3 verbal simple scale

Exclusion Criteria:

1. Personal history of disorders of hemostasis or previous history of abnormal bleeding evidence.
2. Local infection at the site of the puncture or to puncture prior systemic.
3. Contraindications to study medication.
4. Muscle or neurological disease, peripheral or central.
5. Patients with prior history of opioid.
6. Pregnancy or lactation.
7. Difficulties in assessing pain or inability to understand or assist in the development of the study (psychiatric illness, cognitive impairments)
8. Active Chronic alcoholism or drug addiction.
9. BMI under 20 or mayor 30.
10. Chronic treatment with non-steroidal anti-inflammatory drugs, antidepressants, anticonvulsants or opioids.
11. Rejection of the patient

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-09; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
pain score: verbal simple scale | 0,3,6,12,18 and 24h
  admission to post-anesthesia care unit (PACU)
pain score: visual number scale | 0, 3, 6,12, 18, 24h
  post-admission to PACU
opioid requirements | 24 h
  0 dose/ 1 dose/ 2 or more doses
sleep quality | 24 h
  bad/regular/good
amount of sleep | 24 h
  < 3h/ 3-6h, >6h

SECONDARY OUTCOMES:
percentage of participants with nausea and vomiting | 24 hours
  without symptoms/ nausea/vomiting/ both symptoms
Number of Participants with Serious and Non-Serious Adverse Events | 24 h
  directly due to block nerve and general complications

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Abente y Lago. Complejo Hospitalario Universitario A Coruña, A Coruña, Spain